CLINICAL TRIAL: NCT05516056
Title: Enhanced Recovery After Surgery Program in a Low and Middle-income Country: Feasibility, Safety, Patient's Acceptance, Reduction of the Length of Hospital Stay, Bed Turnover and Cost Benefits for Laparoscopic Cholecystectomy at CHUK
Brief Title: ERAS After Cholecystectomy in Kigali, Rwanda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olivier Detry MD PhD (Other)
Collaborators: University of Rwanda (Other)
Responsible Party: Sponsor-Investigator, Olivier Detry MD PhD, Chargé de Cours (Associate Professor), University of Liege
Organization: University of Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/CHUK/074/2021
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: ERAS; Gall Bladder Disease
Keywords: laparoscopy; surgery; Patient oriented outcomes; pain; complication; cholecystectomy; anesthesiology
MeSH Terms: conditions — Gallbladder Diseases; Pain

STUDY DESIGN:
Intervention Model Description: prospective and cross sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERAS group (Experimental): First 50 patients included in the ERAS pathway for cholecystectomy in CHUK, Rwanda
  Interventions: Other: ERAS clinical pathway

INTERVENTIONS:
Other: ERAS clinical pathway — Prospective evaluation of the clinical results of ERAS implementation in the first 50 patients undergoing ERAS for cholecystectomy in CHUK, Rwanda

SUMMARY:
Enhanced Recovery After Surgery (ERAS) pathway represents a peri-operative multimodal management aiming at a decrease in surgical aggression and an improved patient rehabilitation, in order to reduce postoperative morbidity, length of hospital stay and, as an important secondary consequence, overall costs. ERAS pathways have been successfully implemented in many surgical managements in the Western world, but very few data exist on ERAS in developing countries. This project aims at the prospective evaluation of ERAS pathway implementation in cholecystectomies in CHUK, Rwanda. The first 50 patients will be prospectively evaluated and compared to the last 50 patients who underwent cholecystectomy before ERAS pathway implementation.

DETAILED DESCRIPTION:
All adult patients scheduled for laparoscopic cholecystectomy at the CHUK and accepting to be included in the study and the ERAS protocol, will be informed of all steps of the ERAS pathway. Education and discharge plan will be discussed.

A regular ERAS pathway will be proposed. All patients will be allowed to take a regular diet until 6h and carbohydrate loading or clear fluids until 2h before surgery. Thromboembolism prophylaxis with low molecular weight heparins will be administered according to patient's comorbidities. No premedication will be administered. Combined anesthesia technique will be used: general anesthesia added to local infiltration of the surgical incision. In all cases restricted intra-operative fluid administration (6-8 ml/kg/h) and prevention of hypothermia will be used during the procedure. Moreover, no opioids will be used during the whole perioperative period. Antibiotic prophylaxis will be given in agreement with the hospital protocol. Analgesia and prevention of nausea will be given. Immediate postoperative monitoring will be performed in the recovery room where the pain numeric rating scale (NRS) will be routinely evaluated by the anesthesiologist or the NPA.

Laparoscopic approach with a 4-trocar technique will be the first choice when not contraindicated. No abdominal drainage, no nasogastric tube will be used, but, if necessary, it will be placed immediately during or after anesthesia and removed upon awakening. A bladder catheter will be placed if indicated and removed immediately after surgery.

The ERAS anesthesia postoperative care will include: intravenous paracetamol or ketamine administration when necessary, avoidance of opioids, treatment of nausea and vomiting when necessary. Pain will be assessed every 4 h using NRS pain scale by nursing staff, and paracetamol + NSAID will be given if needed.

Re-feeding will be authorized 2h to 4h after surgery with liquid diet and mobilization. Withdrawal of intravenous infusions will be performed at 6h post-operatively. Patient mobilization will be further encouraged and increased gradually. All meals will be consumed sitting at the table. At 24h after surgery, blood tests (FBC and CRP) will be performed and discharge authorized in case of normal vital signs and blood tests, absence of complications or symptoms, digestive function enabling the patient to eat without nausea or vomiting, return of intestinal transit with emission of gas (stool not required), autonomy to move and post-operative pain relief with oral analgesics. The patient will be given oral analgesia for at least 48 hours. After discharge, the surgical team will make follow-up controls by phone on day 3, 5, and 7, to detect any sign of complications during the first week. If no complaint, the outpatient clinic evaluation will be planned at postoperative 15 and 30. A last follow-up control will be performed by phone at day 90.

Data will be collected for age, gender, indications for surgery, American Society of Anesthesiology (ASA) class, operative time, adverse events (pain, nausea and vomiting), length of hospitalization, and intra- and post-operative complications. The expenses of surgery and in-hospital care will be calculated and analyzed. After discharge, on days 3, 10, 15, 30, and 90, patients will report outcomes that will be recorded by Surgical Recovery Scale (SRS).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing scheduled elective laparoscopic cholecystectomy in CHUK, Rwanda
* Signed informed consent

Exclusion Criteria:

* acute cholecystitis
* ASA IV patients
* absence of consent

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From the day of the laparoscopic cholecystectomy to postoperative day 90
  Number of days of hospitalization after laparoscopic cholecystectomy (in days)
Rate of Postoperative complications | From the day of the laparoscopic cholecystectomy to postoperative day 90
  All postoperative complications reported according to the Dindo-Clavien grading of surgical complications, graded from grade 0 (no complication) to death (worst outcome) as grade V. This is the standard grading of surgical complication.

SECONDARY OUTCOMES:
Cost of laparoscopic cholecystectomy | From the day of the laparoscopic cholecystectomy to postoperative day 90
  Total cost of hospitalization and readmission (in Rwandese francs and US $)
Patient satisfaction measured with the Satisfaction Likert Scale (SLS) | From the day of the laparoscopic cholecystectomy to postoperative day 90
  Patient satisfaction measured with the 5-point Satisfaction Likert Scale (1: very dissatisfied; 2: dissatisfied; 3: neutral; 4: satisfied; 5: very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Detry, MD PhD, Principal Investigator — University of Liege
Locations (1):
- Centre Hospitalier Universitaire de Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyundo M, Kayondo K, Gasakure M, Twagirumukiza JD, Gashegu J, Detry O. Implementation and outcomes of an enhanced recovery after surgery pathway for laparoscopic cholecystectomy in East and Central Africa: A prospective non-randomized controlled trial in Rwanda's Tertiary Teaching Hospital. World J Surg. 2025 Mar;49(3):605-614. doi: 10.1002/wjs.12371. Epub 2024 Oct 10. PMID 39390308

DOCUMENTS (2):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT05516056/Prot_000.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT05516056/ICF_001.pdf